CLINICAL TRIAL: NCT02254746
Title: A Phase I-II Dose Escalation Study of Stereotactic Body Radiation Therapy in Patients With Localized Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Dr Fernanda Herrera, Cheffe de clinique, Centre Hospitalier Universitaire Vaudois
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUV-DO-HYPORT-2013
Record Dates: First submitted 2014-09-16; First posted 2014-10-02 (Estimated); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Prostate Adenocarcinoma
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Phase I (dose escalation)/ Phase II (Experimental): Phase I
  * Prostate tumor: starting dose 9 Gy per fraction in 5 fractions (total 45 Gy) and subsequent dose escalation up to 10 Gy.
  * Prostate gland: fixed prophylactic tumoricidal dose 7.25 Gy per fraction in 5 fractions (no dose escalation). Total 36.25 Gy.
  Phase II
  Additional patients will be treated at either the maximum tolerated dose (MTD) or at the highest dose level as determined by the investigators from the Phase I portion of the study.
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy (SBRT)

SUMMARY:
The aim of this study is to test the safety and efficacy of Stereotactic Body Radiation Therapy (SBRT) in localized prostate carcinoma in patients for whom the standard treatment is the irradiation of the entire prostate gland with or without seminal vesicles accompanied or not by hormonal therapy. In light of the accumulating clinical evidence favoring the use of hypo fractionation, SBRT regimen might constitute a much more convenient non-invasive and highly efficient outpatient therapy.

DETAILED DESCRIPTION:
Primary objective phase I:

To irradiate the prostate gland which might albeit contain microscopic disease with tumoricidal doses of SBRT, and to escalate the dose of SBRT in the visible prostatic tumor towards the best tumoricidal dose without exceeding the normal tissue tolerance and toxicity in patients with organ confined T2-T3 N0 prostate carcinoma.

Primary objective phase II:

To determine the rate of acute toxicity grade 2 or more defined as toxicity occurring immediately after the first fraction of radiotherapy and up to 90 days after the start of radiotherapy treatment.

Secondary objectives phase II:

* To determine efficacy measured by PSA failure using Phoenix definition.
* To determine long-term late toxicity (>90 days after treatment start).

Exploratory endpoint phase II:

• To determine the feasibility of achieving dose constraints in the organs at risk using high technology radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* All patients must be willing and capable to provide informed consent
* Histologic confirmation of prostate adenocarcinoma
* T2-T3 tumors, N0 (clinically by no evidence of metastatic lymph nodes on CT or MRI)
* No direct evidence of regional or distant metastases
* PSA less than or equal to 50 μg/ml
* Visible gross tumor at the prostate endorectal coil MRI.
* The ultrasound or MRI based volume estimation of the patient's prostate gland no greater than 70g or 70cc
* No significant urinary obstructive symptoms; IPSS score must be ≤ 15 (alpha blockers allowed)
* Patient must have undergone an endorectal coil magnetic resonance image (MRI) of the prostatic gland (before rectal spacer if any),
* Patient must have undergone the following assessments in case of PSA ≥ 20μg/L, and/or T3 tumor and/or Gleason Score ≥ 8:

  * bone scan
  * Chest abdominal and pelvis computed tomography (CT) scan
* If tumor is localized at less than 3 mm from the rectum a rectal spacer is mandatory. Patient accepts the rectal spacer to be injected before treatment starts
* Patient accepts to have one planning MRI after the injection of rectal spacer (without endorectal coil)
* Patient accepts the preparation of the bladder (bladder full), before the planning MRI, planning CT and then before each treatment fraction

Exclusion Criteria:

* Previous radiotherapy in the pelvis
* Tumor localized at less than 3 mm from the urethra
* History of inflammatory colitis (including Crohn's disease and ulcerative colitis)
* Prior cancer in the pelvis
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before inclusion in the trial

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2023-11-08 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (phase I) | During the first 30 days from the start of treatment
  Observation of dose-limiting toxicities (DLT) defined as any treatment-related grade ≥ 3 acute toxicity occurring in the radiation field or irradiated volumes in the following categories GI or GU. In addition, any other grade 4 or 5 toxicity attributed to the therapy constitutes a DLT.
Toxicity (phase II) | 90 days after the first fraction of radiotherapy treatment
  Acute GU and GI toxicity (grade 2 or more) according to the NCI CTCAE v4.0.

SECONDARY OUTCOMES:
Efficacy (phase II) | 3 monthly assessments during the first 2 years and 6 monthly assessments until end of study (5 years)
  PSA failure using Phoenix definition
Toxicity (phase II) | > 90 days and up to 5 years from the start of protocol treatment
  Long term GU and GI toxicity (grade 2 or more) according to the NCI CTCAE v4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda Herrera, MD, Principal Investigator — CHUV
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No